CLINICAL TRIAL: NCT05093127
Title: CArotid Robotic Procedure Evaluation
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Robocath (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: ROB-02
Record Dates: First submitted 2021-09-30; First posted 2021-10-26 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Carotid Artery Stenting — R-OneTM system is a tool available to physicians for performing CAS without changing the treatment of the pathology. R-OneTM system is designed to remotely deliver and manipulate guidewires and stent/balloon devices during Carotid Artery Stenting. The system is composed of the R-OneTM robotic platform used in combination with two accessories, the Mobile radioprotection screen and a sterile and single-use R-OneTM consumable kit. The physician, seated at the remote radio-protected control station, manipulates guidewires and/or balloon/stent catheters using joysticks on the Command unit.

SUMMARY:
This study aims to evaluate the use of R-One in the peripheral vasculature.

DETAILED DESCRIPTION:
This is a prospective, single-arm, monocenter study to evaluate the R-one use in carotid artery stenting procedures. Up to 8 patients will be included and followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Candidate for CAS
3. Presence of a WEB-diaphragm lesion at carotid artery ostium, proved by non-invasive imaging (CTA or MRA)
4. No minimum delay between previous stroke therapy (IMT) is required
5. Double antiplatelet therapy the day before the procedure and 1 month after the procedure is required
6. The patient provides written informed consent as approved by the applicable Ethics Committee and is willing to comply with all study requirements including 30 days follow-up.
7. The patient is affiliated with a social security scheme

Exclusion Criteria:

1. Target lesion has atherosclerotic or dissection stenosis or occlusion;
2. Treatment of in-stent restenosis, or prior stent in the target vessel proximal to the target lesion;
3. CAS performed at the end of intracranial mechanical thrombectomy
4. Contra-indications of double antiplatelet therapy the day before the procedure and 1 month after the procedure
5. Patients under judicial protection, tutorship or curatorship
6. Any patient participating in another clinical study valuating a drug or a medical device (except registries for which the primary endpoint has not been evaluated);
7. Pregnant and breast-feeding women or intention to become pregnant prior to completion of all follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 8 Patients with carotid artery disease, including patients with web diaphragm, who qualify for Carotid Artery Stenting.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Procedure technical success | Index Procedure : Day 0
  Absence of any unplanned manual assistance or conversion to manual CAS for procedural completion

SECONDARY OUTCOMES:
Absence of intra-procedural complications | At Day 0 and at Day 30 +/- 7 days
  Absence of major stroke which required intracranial mechanical thrombectomy or IV-thrombolysis, perforation of carotid artery, acute occlusion of carotid artery or significant thrombus formation, significant air embolus during the procedure.
Reduction in primary operator radiation exposure | Index Procedure : At Day 0
  Reduction of Primary Operator Radiation Exposure measured by dedicated dosimeters, defined as the ratio of the radiation dose measured at the primary operator during the overall procedure to the radiation exposure measured at the procedure table (the conventional site of the primary operator during the procedure).
Radiation exposure for the patient | Index Procedure: At Day 0
  Dose measured by the imaging system during the procedure.
Overall Procedure Time | Index Procedure : At Day 0
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Overall contrast volume | Index Procedure : At Day 0
  Total volume of contrast (mL) used during the procedure.
Contrast volume during Robotic Procedure | Index Procedure : At Day 0
  Total volume of contrast (mL) used during the robotic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: François EUGENE, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Hôpital Pontchaillou - CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided